CLINICAL TRIAL: NCT07303907
Title: An Open-label Study Evaluating MM402 in Adults With Autism Spectrum Disorder
Brief Title: A Phase 2A Trial of MM402 for Autism Spectrum Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Definium Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM402-105
Record Dates: First submitted 2025-12-22; First posted 2025-12-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; ASD
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 200 mg MM402 (R-MDMA) (Experimental): A psychoactive substance that mediates effects mainly through a release of the monoaminergic neurotransmitters, with the greatest effect on 5-HT, followed by NE and DA
  Interventions: Drug: MM402 (R-enantiomer of 3,4-methylenedioxymethamphetamine (MDMA))

INTERVENTIONS:
Drug: MM402 (R-enantiomer of 3,4-methylenedioxymethamphetamine (MDMA)) — A psychoactive substance that mediates effects mainly through a release of the monoaminergic neurotransmitters, with the greatest effect on 5-HT, followed by NE and DA
  Other Names: MDMA

SUMMARY:
A Phase 2A Trial of MM402 Open-Label Study in Adults with Autism Spectrum Disorder

DETAILED DESCRIPTION:
This study will enroll approximately twenty adults with Autism Spectrum Disorder (ASD) aged 18 to 45 years of age.

This is a single-center, open-label study to evaluate the effects after a single administration of MM402 to adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ASD per records as confirmed by standard semi-structured interview for Autism diagnosis (eg, Autism Diagnostic Observation Schedule-Second Edition)
2. Male or Female aged 18 to 45
3. Presents with clinically significant deficits in socialization and communication as determined by Social Responsiveness Scales (SRS-2) ≥66

Exclusion Criteria:

1. Has uncorrected abnormalities in eye movement, alignment, or acuity or atypical eye features that could interfere with eye tracking
2. First degree relative with or lifetime history of a psychotic disorder or bipolar disorder
3. Current diagnosis of alcohol or substance use disorder (excluding nicotine and caffeine)
4. Any clinically significant unstable illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 11-point Numerical Rating Scale (NRS) scores | Baseline, pre-dose and 2, 4, 6, 8, and 24 hours post-dose and day 15
  The NRS is an 11-point PRO scale used to measure the severity or intensity of effects from 0 (no effect) to 10 (high severity or intensity of effect). It consists of various items related to both positive and negative effects in the autism patient population.

SECONDARY OUTCOMES:
Subjective 5-question Drug Effects Questionnaire (DEQ) scores | 1, 2, 4, 6, 8, and 24 hours post-dose
  The Drug Effects Questionnaire is used in studies to assess the participant's acute subjective effects after ingesting substances. It consists of 5 PRO items. The analog scale of responses ranges from "not at all" to "extremely." The score is determined by the distance between the left anchor point and the participant's mark on the line. Each item is scored separately.
Pharmacokinetic Plasma concentrations | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Maximum Plasma Concentration [Cmax] of MM402 in the blood.
Pharmacokinetic Parameters (Cmax) | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Maximum concentration (Cmax).
Pharmacokinetic Parameters (Tmax) | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Time to maximum concentration (Tmax).
Pharmacokinetic Parameters (t1/2) | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Time to maximum concentration half-life (t1/2).
Pharmacokinetic Parameters (AUC0-inf) | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Area under the concentration curve from time 0 to infinity (AUC0-inf).
Pharmacokinetic Parameters (AUC0-24h) | pre-dose and 1, 2, 4, 6, 8, and 24 hours post-dose
  Area under the concentration curve from time 0 to 24 hour (AUC0-24h).

CONTACTS AND LOCATIONS:
Locations (1):
- Spectrum Neuroscience and Treatment Institute, New York, New York, United States